CLINICAL TRIAL: NCT00553774
Title: Effect of Cocoa Flavanols on Vascular Function in Optimally Treated Coronary Artery Disease Patients: Interaction Between Endothelial Progenitor Cells, Reactivity of Micro- and Macrocirculation
Brief Title: Effect of Cocoa Flavanols on Vascular Function
Acronym: Cocoa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Yerem Yeghiazarians, Proffessor of Clinical Medicine, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CHR#H47369-28112
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease
Keywords: CAD Patients on Optimal Treatment
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flavanol (Experimental): Cocoa Flavanol
  Interventions: Dietary Supplement: Cocoa Flavanols
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cocoa Flavanols — Cocoa Flavanols (BD for 21 - 28 days)
  Arms: Flavanol
Other: Placebo — Placebo (BD 21 - 28 Days)
  Arms: Placebo

SUMMARY:
Endothelial dysfunction is associated with a higher incidence of adverse cardiovascular events in patients with coronary artery disease (CAD). CAD patients also show impaired function and number of endothelial progenitor cells (EPCs, adult stem cells) which circulate in adult blood and contribute to endothelial repair. Clinical studies suggest that endothelial function can be improved in CAD patients by consumption of flavanol-rich cocoa. Yet, the mechanism is not known. It is also not known whether flavanol-rich cocoa provides an additive, positive effect in patients who are already receiving the maximal recommended therapies for risk factor modification. Therefore, the researchers propose to perform an investigator-initiated, randomized controlled cross-over study administering flavanol-rich cocoa or a placebo for two months in CAD patients on optimal medical therapy. An improvement of endothelial function as measured by flow-mediated dilation (FMD) will be the primary endpoint of this study. The researchers propose to also measure determinants of FMD such as microvascular response, inflammatory markers, metabolites of nitric oxide, as well as the number and function of EPCs in the blood. Importantly, detailed food questionnaires and plasma flavanols/metabolites will help to further support a causal link between flavanol-intake and improved vascular function.

ELIGIBILITY:
Inclusion Criteria:

* CAD patients over 18 years of age
* Contact university for more details.

Exclusion Criteria:

* Contact university for more details.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
An improvement of endothelial function as measured by flow-mediated dilation (FMD) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Yerem Yeghiazarians, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

REFERENCES:
- [Derived] Heiss C, Jahn S, Taylor M, Real WM, Angeli FS, Wong ML, Amabile N, Prasad M, Rassaf T, Ottaviani JI, Mihardja S, Keen CL, Springer ML, Boyle A, Grossman W, Glantz SA, Schroeter H, Yeghiazarians Y. Improvement of endothelial function with dietary flavanols is associated with mobilization of circulating angiogenic cells in patients with coronary artery disease. J Am Coll Cardiol. 2010 Jul 13;56(3):218-24. doi: 10.1016/j.jacc.2010.03.039. PMID 20620742